CLINICAL TRIAL: NCT01190111
Title: An Open-label, Multicenter Study of Subcutaneous Intermittent Recombinant Interleukin-7 (CYT107) in Chronically HIV-infected Patients With CD4 T-lymphocyte Counts Between 101-400 Cells/mm3 and Plasma HIV RNA< 50 Copies/mL After at Least 12 Months of HAART
Brief Title: Study on Interleukin-7 (CYT107) in HIV Patients
Acronym: Inspire 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CYTHERISSA filed for banckcuptcy in June 2013.Subjects treated by CYT 107 were followed up for at the least 3 months.
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-13
Record Dates: First submitted 2010-08-23; First posted 2010-08-27 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: HIV
Keywords: interleukin-7; immune-based therapy; HIV; viral disease
MeSH Terms: conditions — Virus Diseases | interventions — Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYT107 (r-hIL-7) (Experimental)
  Interventions: Biological: Interleukin-7

INTERVENTIONS:
Biological: Interleukin-7 — 20 µg/kg/week. 3 administrations, 1 per week (1 cycle) repeated cycles based on a CD4-guided response
  Other Names: CYT107

SUMMARY:
This study was designed to evaluate the pharmacokinetics of 20µg/kg/week of Interleukin-7 (CYT107), the biological activity and safety of repeated cycles of CYT107, for a maximum of 4 cycles within 21 months and a maximum of 3 cycles within 12 months.

DETAILED DESCRIPTION:
This was a phase IIa study assessing weekly doses of CYT107 in addition to antiviral treatment (HAART) in adult patients with HIV.

CYT107 were administered at the dose of 20 µg/kg based on the patient's weight, in 3 weekly administrations. CYT107 Subcutaneous injection administered at the clinic or day hospital

Patients were followed every 3 months for primary and secondary biological activity criteria as well as safety up to 24 months long term follow-up with quarterly visits.

A cycle = 3 weekly administrations; D/d0; D/d7; D/d14 For all patients there will be a maximum of 3 cycles over 12 months and a maximum of 4 cycles over 21 months, for a total duration on study of 24 months.

All patients were receiving and continued to receive combination antiretroviral therapy while on-study.

Pre-medication was not be used systematically but might be administered if needed according to standard clinical practice.

During the study visits the following may be done:

* Medical history, physical examination, blood tests every visit.
* Electrocardiogram (EKG)
* Chest x-ray study
* Liver/spleen imaging
* Blood sample collections at frequent intervals for laboratory tests (Virology: HIV RNA &HIV DNA;Pharmacodynamics/Immunology;Bacterial translocation )
* Urine tests several times during the study.

PBMCs collections for immunological testing

An optional substudy on gut biopsy performed prior and at month 3 after the first CYT107 cycle to evaluate T cell homing

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western Blot at any time prior to study entry.
* Age ≥18.
* On HAART for at least 12 months, on stable regimen for at least 3 months prior to enrollment. HAART is defined as a combination of 2 classes dose regimen of approved ARV.
* CD4 cell counts ≥ 101 and < 400 cells/mm3 on two (2) consecutive measurements (including the screening value) within the previous 12 months prior to enrollment.
* Plasma HIV RNA < 50 copies/mL on at least two consecutive measurements (including the screening value) within the previous 6 months prior to enrollment. Note: Patients with single blip of detectable viremia during this period (6 months prior screening) will be allowed to participate if the prior and subsequent plasma HIV RNA levels are below the limits of detection.
* No AIDS-defining illness (category C) diagnosed within the last 6 months prior to enrollment.

Exclusion Criteria:

* Use of any other investigational antiretroviral agents.
* Any planned or probable modification of the anti-retroviral treatment during the first 3 month study period.
* Current or recent history (<30 days prior to screening) of a viral, bacterial, parasitic or fungal infection requiring systemic treatment and/or hospitalization.
* Positive PPD unless there is documentation of completion of INH therapy for latent tuberculosis.
* Any serious illness requiring systemic treatment and/or hospitalization until the patient either completes therapy or is clinically stable on therapy, in the opinion of the principal investigator, for at least 28 days prior to study .
* Any history of malignancy (except basal carcinoma of the skin) including any hematologic malignancy or AIDS defining malignancy, such as lymphoproliferative disorder or Kaposi's sarcoma. (Patients with Kaposi's sarcoma limited to the skin that disappeared while on HAART therapy, and without requiring any other systemic therapy, 1 year prior to study entry will be eligible to participate).
* Any history of HIV related encephalopathy.
* Hepatitis B or C (positive HBs Ag or positive anti HBc antibodies with a detectable HBV DNA viral load or positive anti HCV antibodies with a detectable HCV RNA viral load). Patients who became negative to HBV DNA or HCV RNA following an antiviral treatment should not be enrolled.
* HIV-2, HTLV-1 or HTLV-2 seropositivity.
* Pregnant or lactating women. Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week prior to study entry.
* Refusal or inability to practice contraception regardless of the gender of the patient.
* Hypertension with a resting systolic blood pressure > 140 or a resting diastolic blood pressure > 90 mm despite adequate antihypertensive treatment.
* Use of tipranavir/ritonavir (TPV/r) and Enfuvirtide (T-20).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
• To study, in all included patients, the biological activity and safety of repeated cycles of CYT107, for a maximum of 4 cycles within 21 months and a maximum of 3 cycles within 12 months. | 2 years (24 months)

SECONDARY OUTCOMES:
• To characterize in the first 12 patients, PK and PD of CYT107 . • To further characterize in all included patients, the safety profile established with CYT107 at 20 µg/kg including monitoring of HIV RNA and immunogenicity. • • • | 2 years
  * To characterize in the first 12 patients, PK and PD of CYT107 .
  * To further characterize, the safety profile established with CYT107 at 20 µg/kg including monitoring of HIV RNA and immunogenicity.
  * To further examine CYT107 effect on HIV specific T-cells.
  * To document other properties of IL-7, (ie: T-cell homing within the GI tract).
  * To assess the sustained CD4 increase until the end of the two years
    * the safety of CYT107 treatment over the same period
    * the potential effect of the CYT107 induced immune reconstitution on HIV-induced chronic systemic immune hyper-activation and its consequences

OTHER OUTCOMES:
clinical and lab assessment Imaging, EKG and Ultrasound IL-7 Pharmacokinetics and Immunogenicity IL-7 Pharmacodynamics/Immunology Bacterial Translocation and HLA typing | every 3 months up to the end of study period 2years
  Immune Monitoring will consist on T-cell subsets identification and quantification (such as RTE, naïve/effector and memory CD4 and CD8 T-cells, B cells, CD4 CD25 Fox P3 regulatory T-cells), quantification of the expression of CD127 and the evaluation of T-cell cycling and survival.
  T-cell Repertoire Diversity:
  Thymopoiesis Evaluation: Quantification of sjTRECs and βTRECs will be done by Real Time Quantitative PCR, and Ratio values will be analyzed.
  GUT Biopsy - T-cell Homing :Essential receptors expression for intestinal homing, namely the integrin α4β7 and CCR9, the receptor for the gut-associated chemokine TECK/CCL25 could be assessed as well as molecules for T-cell trafficking (CCR7, CXCR4, CXCL12...) in the gut biopsies.
  Immunogenicity: antidrug antibody (ADA) and neutralizing ADA will be tested. In case of a positive sample, the test will be repeated every 3 months until negative.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Lederman,, Pr, Study Chair — Case Western Reserve University
Locations (4):
- United States (3):
  - University of Miami School of Medicine, Miami, Florida
  - Niaid/Nih, Bethesda, Maryland
  - Case Western Reserve University, Cleveland, Ohio
- McGill University Health Center (MUHC), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Thiebaut R, Jarne A, Routy JP, Sereti I, Fischl M, Ive P, Speck RF, D'Offizi G, Casari S, Commenges D, Foulkes S, Natarajan V, Croughs T, Delfraissy JF, Tambussi G, Levy Y, Lederman MM. Repeated Cycles of Recombinant Human Interleukin 7 in HIV-Infected Patients With Low CD4 T-Cell Reconstitution on Antiretroviral Therapy: Results of 2 Phase II Multicenter Studies. Clin Infect Dis. 2016 May 1;62(9):1178-1185. doi: 10.1093/cid/ciw065. Epub 2016 Feb 7. PMID 26908786